CLINICAL TRIAL: NCT04901871
Title: ED50 and ED95 of Remimazolam Intravenous Bolus on the Loss of Consciousness in Patients Undergoing General Anesthesia
Brief Title: Remimazolam Bolus for General Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Woo Han, Associate professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 3-2021-0091
Record Dates: First submitted 2021-05-10; First posted 2021-05-26 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Loss of Consciousness
MeSH Terms: conditions — Unconsciousness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- 1 (0.02 mg/kg, age<65) (Active Comparator): Remimazolam of 0.02 mg/kg will be infused in patients aged<65.
  Interventions: Drug: 0.02 mg/kg, age<65
- 2 (0.07 mg/kg, age<65) (Active Comparator): Remimazolam of 0.07 mg/kg will be infused in patients aged<65.
  Interventions: Drug: 0.07 mg/kg, age<65
- 3 (0.12 mg/kg, age<65) (Active Comparator): Remimazolam of 0.12 mg/kg will be infused in patients aged<65.
  Interventions: Drug: 0.12 mg/kg, age<65
- 4 (0.17 mg/kg, age<65) (Active Comparator): Remimazolam of 0.17 mg/kg will be infused in patients aged<65.
  Interventions: Drug: 0.17 mg/kg, age<65
- 5(0.22 mg/kg, age<65) (Active Comparator): Remimazolam of 0.22 mg/kg will be infused in patients aged<65.
  Interventions: Drug: 0.22 mg/kg, age<65
- 6(0.27 mg/kg, age<65) (Active Comparator): Remimazolam of 0.27 mg/kg will be infused in patients aged<65.
  Interventions: Drug: 0.27 mg/kg, age<65
- 7 (0.02 mg/kg, age≥65) (Active Comparator): Remimazolam of 0.02 mg/kg will be infused in patients aged≥65.
  Interventions: Drug: 0.02 mg/kg, age≥65
- 8 (0.07 mg/kg, age≥65) (Active Comparator): Remimazolam of 0.07 mg/kg will be infused in patients aged≥65.
  Interventions: Drug: 0.07 mg/kg, age≥65
- 9 (0.12 mg/kg, age≥65) (Active Comparator): Remimazolam of 0.12 mg/kg will be infused in patients aged≥65.
  Interventions: Drug: 0.12 mg/kg, age≥65
- 10 (0.17 mg/kg, age≥65) (Active Comparator): Remimazolam of 0.17 mg/kg will be infused in patients aged≥65.
  Interventions: Drug: 0.17 mg/kg, age≥65
- 11 (0.22 mg/kg, age≥65) (Active Comparator): Remimazolam of 0.22 mg/kg will be infused in patients aged≥65.
  Interventions: Drug: 0.22 mg/kg, age≥65
- 12 (0.27 mg/kg, age≥65) (Active Comparator): Remimazolam of 0.27 mg/kg will be infused in patients aged≥65.
  Interventions: Drug: 0.27 mg/kg, age≥65

INTERVENTIONS:
Drug: 0.02 mg/kg, age<65 — Remimazolam of 0.02 mg/kg will be infused in patients aged<65.
  Arms: 1 (0.02 mg/kg, age<65)
Drug: 0.07 mg/kg, age<65 — Remimazolam of 0.07 mg/kg will be infused in patients aged<65.
  Arms: 2 (0.07 mg/kg, age<65)
Drug: 0.12 mg/kg, age<65 — Remimazolam of 0.12 mg/kg will be infused in patients aged<65.
  Arms: 3 (0.12 mg/kg, age<65)
Drug: 0.17 mg/kg, age<65 — Remimazolam of 0.17 mg/kg will be infused in patients aged<65.
  Arms: 4 (0.17 mg/kg, age<65)
Drug: 0.22 mg/kg, age<65 — Remimazolam of 0.22 mg/kg will be infused in patients aged<65.
  Arms: 5(0.22 mg/kg, age<65)
Drug: 0.27 mg/kg, age<65 — Remimazolam of 0.27 mg/kg will be infused in patients aged<65.
  Arms: 6(0.27 mg/kg, age<65)
Drug: 0.02 mg/kg, age≥65 — Remimazolam of 0.02 mg/kg will be infused in patients aged≥65.
  Arms: 7 (0.02 mg/kg, age≥65)
Drug: 0.07 mg/kg, age≥65 — Remimazolam of 0.07 mg/kg will be infused in patients aged≥65.
  Arms: 8 (0.07 mg/kg, age≥65)
Drug: 0.12 mg/kg, age≥65 — Remimazolam of 0.12 mg/kg will be infused in patients aged≥65
  Arms: 9 (0.12 mg/kg, age≥65)
Drug: 0.17 mg/kg, age≥65 — Remimazolam of 0.17 mg/kg will be infused in patients aged≥65.
  Arms: 10 (0.17 mg/kg, age≥65)
Drug: 0.22 mg/kg, age≥65 — Remimazolam of 0.22 mg/kg will be infused in patients aged≥65.
  Arms: 11 (0.22 mg/kg, age≥65)
Drug: 0.27 mg/kg, age≥65 — Remimazolam of 0.27 mg/kg will be infused in patients aged≥65.
  Arms: 12 (0.27 mg/kg, age≥65)

SUMMARY:
It is important to estimate the adequate dose of remimazolam intravenous bolus injection to induce the loss of consciousness. We will determine the ED50 and ED95 of remimazolam intravenous bolus on the loss of consciousness in patients undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years old or older, with American Society of Anesthesiologists Physical Status 1-3, and scheduled for general anesthesia

Exclusion Criteria:

1. Patients scheduled for liver surgery
2. Uncontrolled hypertension
3. Uncontrolled diabetes mellitus
4. Liver disease
5. Kidney disease
6. Intolerance or hypersensitivity to benzodiazepine
7. Addiction
8. Glaucoma
9. Heart failure
10. Peripheral vascular disease
11. Obstuctive lung disease
12. Patients scheduled for regional anesthesia before general anesthesia
13. Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Loss of consciousness within 5 minutes | At 5 minutes after infusion
  Loss of consciousness will be evaluated at 5 minutes after infusion.

SECONDARY OUTCOMES:
Time to loss of consciousness | At 5 minutes after infusion (time to loss of consciousness)
  Time to loss of consciousness will be assessed at 5 minutes after infusion.
blood pressure | At 5 minutes after infusion
  Blood pressure will be measured at 0, 1, 2, 3, 4, 5 minutes after infusion.
heart rate | At 5 minutes after infusion
  Heart rate will be measured at 0, 1, 2, 3, 4, 5 minutes after infusion.
sedline | At 5 minutes after infusion
  Sedline will be measured at 0, 1, 2, 3, 4, 5 minutes after infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Woo Han, Principal Investigator — GangnamSeveracne Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Chae D, Kim HC, Song Y, Choi YS, Han DW. Pharmacodynamic analysis of intravenous bolus remimazolam for loss of consciousness in patients undergoing general anaesthesia: a randomised, prospective, double-blind study. Br J Anaesth. 2022 Jul;129(1):49-57. doi: 10.1016/j.bja.2022.02.040. Epub 2022 May 11. PMID 35562226